CLINICAL TRIAL: NCT02291276
Title: Perioperative Assessment of Right Ventricular Function and Venous Return in Patients With Epithelial Ovarian Cancer Undergoing Cytoreductive Surgery (GynRight) - Pilot Study
Brief Title: Perioperative Assessment of Right Ventricular Function and Venous Return in Patients With Epithelial Ovarian Cancer Undergoing Cytoreductive Surgery (Gyn Right) - Pilot Study
Status: Withdrawn | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Claudia Spies, Univ.- Prof. Dr. Claudia Spies, Charite University, Berlin, Germany
Other Study IDs: GynRight
Record Dates: First submitted 2014-11-07; First posted 2014-11-14 (Estimated); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Right Ventricular Function and Venous Return

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Female cancer patients with ascites: Primary epithelial ovarian female cancer patients with ascites (> 500 ml ascites in the preoperative sonographic examination)
- Female cancer patients aged > 70 years: Primary epithelial ovarian female cancer patients aged > 70 years with at least one of the following secondary diagnoses:
  * Status Post stent placement due to coronary heart disease respectively Status Post-myocardial infarction
  * existing arterial Hypertension for more than 5 years
  * chronic heart failure (New York Heart Association (NYHA) class II-III)
  * peripheral arterial disease

SUMMARY:
In this prospective, observational study the investigators assess the perioperative course of right ventricular function in combination with the venous return in patients undergoing major non-cardiac surgery. The study aims to investigate if patients undergoing major non-cardiac surgery develop an impairment of right ventricular function and/or venous return. Furthermore, the study evaluates if an impairment of right ventricular function and/or venous return is associated to left ventricular function, arterial side of the circulation and to postoperative clinical outcome.

ELIGIBILITY:
Inclusion Criteria:

* Offered patient information and written informed consent
* Female patients aged greater than or equal to 18 years for cytoreductive surgery of a primary epithelial ovarian tumour

  1. Patient Group 1: Female patients with > 500 ml ascites in the preoperative sonographic examination
  2. Patient group 2: Female patients aged > 70 years and at least one of the following secondary diagnoses:

     * Status Post stent placement due to coronary heart disease respectively Status Post-myocardial infarction
     * existing arterial Hypertension for more than 5 years
     * chronic heart failure (New York Heart Association (NYHA) class II-III)
     * peripheral arterial disease

Exclusion Criteria:

* Patients aged less than 18 years
* Persons without the capacity to consent
* Inability of German language use
* Lacking willingness to save and hand out data within the study
* Accommodation in an institution due to an official or judicial order
* (Unclear) history of alcohol or substances disabuse
* Coworker of the Charité
* Advanced disease of the oesophagus or upper respiratory tract at the beginning of hospitalization
* Operation in the area of the oesophagus or nasopharynx within the last two months before participation in the study
* Neurological or psychiatric disease at the beginning of hospitalization
* CHF (congestive heart failure) according to (New York Heart Association) classification - NYHA class IV at the beginning of hospitalization
* American Society of Anesthesiologists (ASA) classification greater than IV
* Renal insufficiency (dependency of haemodialysis) at the beginning of hospitalization
* Pulmonary oedema in thorax x-ray at the beginning of hospitalization
* History of intracranial hemorrhage within one year before participation in the study
* Conditions following venous thrombosis within the last three years before study inclusion
* Known allergies or hypersensitivity on colloidal, starch or gelatine infusion solutions
* Diabetes mellitus with signs of severe neuropathy
* Known atrial fibrillation
* Participation in an interventional clinical trial during the study period; exception: assignment to adjuvant therapy study during this study is allowed.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female cancer patients being observed in the Department of Anesthesiology and Intensive Care Medicine CVK and CCM in cooperation with the Department of Gynecology and Obstetrics CVK at the Campus Virchow - Klinikum, Charité - Universitaetsmedizin Berlin
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Right ventricular function | Up to the first postoperative day
  Right ventricular function will be measured perioperatively by a combination of right ventricular stroke volume, tricuspid annular plane systolic excursion (TAPSE), hepatic venous blood flow, variations in diameter of vena cavae, and right ventricle/left ventricle-ratio.
Venous return | Up to the first postoperative day
  Venous return will be assessed perioperatively by venous return pressure gradient (dVR)

SECONDARY OUTCOMES:
Variables of transthoracic and transesophageal echocardiography | Up to the first postoperative day
  Perioperative course of variables of transthoracic and transesophageal echocardiography
Venous return variables according to Guyton concept | Up to the first postoperative day
  Perioperative course of variables according to Guyton concept characterizing venous return
Hemodynamic variables | Up to the third postoperative day
  Hemodynamic variables are assessed by the anesthesia monitor and esophageal Doppler Monitor
Catecholamine administration | Up to the third postoperative day
  Catecholamine administration intra- und postoperative
Immunological parameter | Up to the third postoperative day
  Perioperative immunological (IL-6 und TNF-alpha)
Endothelial parameter | Up to the third postoperative day
  Perioperative endothelial Parameter (ICAM-1)
Microvascular function | Up to the first postoperative day
  Perioperative course of variables assessing microvascular function
Blood loss | Up to the third postoperative day
  Blood loss characteristics intra- und postoperative
Fluid balance | Up to the third postoperative day
  Fluid and volume administration and balance intra- und postoperative
Organ complications | Participants will be followed up until hospital discharge, an average of two weeks
  Postoperative organ complications are classified according to Clavien - Dindo classification
Postoperative pain | Up to the third postoperative day
  Postoperative pain will be measured by Numeric Rating Scale - Visualized (NRS-V), the Faces Pain Scale - Revised (FPS-R), the Behavioral Pain Scale (BPS) or the Behavioral Pain Scale for Non-Intubated (BPS-NI)
Hospital length of stay | Participants will be followed up until hospital discharge, an average of two weeks
Intensive care unit length of stay | Participants will be followed up until intensive crae unit discharge, an average of two days
Quality of life | Baseline and hospital discharge with an expected average of 14 days
  Assessed with EQ-5D questionnaire
Functional status | Baseline and hospital discharge with an expected average stay of 14 days
  Measured by the Barthel activities of daily living (ADL) index and activities of daily living (IADL).

OTHER OUTCOMES:
Evaluation of right ventricular function index | Up to the first postoperative day
  Right ventricular function index will be evaluated by a combination of right ventricular stroke volume, tricuspid annular plane systolic excursion (TAPSE), hepatic venous blood flow, variations in diameter of vena cavae and right ventricle/left ventricle-ratio.

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Spies, MD, Prof., Study Director — Charite University, Berlin, Germany
Locations (1):
- Department of Anesthesiology and Intensive Care Medicine, Campus Virchow Klinikum, Charité - Universitaetsmedizin, Berlin, Germany